CLINICAL TRIAL: NCT07306156
Title: GP350 CAR-T Cells for Relapse/Refractory and Epstein-Barr Virus Infection Associated Lymphoid Neoplasms, an Open-label, Single-arm Clinical Trial
Brief Title: GP350 CAR-T for Relapse/Refractory and Epstein-Barr Virus Infection Associated Lymphoid Neoplasms
Acronym: ANXIN-02
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhimin Zhai (Other)
Collaborators: Zeno Therapeutics Pte. Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Zhimin Zhai, Chief of Hematology Department, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2025-001
Record Dates: First submitted 2025-12-11; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: EBV Associated Lymphoid Neoplasms
Keywords: LAHS; EBV; Lymphoma; Lymphoid neoplasms; CAR-T
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Treatment (Experimental)
  Interventions: Biological: GP350 CAR-T

INTERVENTIONS:
Biological: GP350 CAR-T — Lymphodepletion chemotherapy with ﬂudarabine (25 mg/m²/day) and cyclophosphamide (250 mg/m²/day) should be administered for 2-3 consecutive days, with the final dose completed 48 hours before infusion. Alternatively, investigators may individualize this regimen based on the subject's specific clinical circumstances.
  The target dose of GP350 CAR-T cells is 1.0-5.0×10⁶ CAR-T cells per kilogram of body weight, administered via intravenous injection. (The actual infused dose is allowed to vary within ±20% from the target dose, depending on the as-released product yield)
  Patients with less than partial response AND without > Grade 2 CRS or any ICANS may receive 1 to 2 additional infusion of GP350 CAR-T cells at the same dose.

SUMMARY:
This is a Phase 1/Phase 2 open-label, single-arm clinical study of GP350 CAR-T for Relapse/Refractory and Epstein-Barr virus infection associated lymphoid neoplasms.

Each participant will undergo leukapheresis after enrolment, receive treatment of the conditioning chemotherapy, and an intravenous infusion of CAR-T cells.

Each participant will proceed through the following study procedures:

* Screening
* Enrollment/Leukapheresis
* Conditioning chemotherapy
* CAR T treatment
* Post-treatment assessment
* Long-term follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Confirmed diagnosis of lymphoid neoplasms according to WHO-HAEM5 (Alaggio R. et al. doi:10.1038/s41375-022-01620-2);
2. Disease Assessment:

   1. Criteria for Relapsed/Refractory lymphoid neoplasms: Meeting any one of the following three conditions: ① Failure to achieve at least a partial response (PR) per Lugano criteria after two cycles of standard first-line therapy; ② Disease progression within six months after achieving a response to first-line therapy, or progression after six months with no response to the original first-line or second-line regimen; ③ Relapse after hematopoietic stem cell transplantation.
   2. Criteria for EBV Infection: Meeting any one of the following three conditions: ① Peripheral blood (plasma or whole blood) EBV DNA load ≥ 10³ copies/ml by quantitative PCR; ②Tumor cell GP350 positivity (≥10% of tumor cells by immunohistochemistry or flow cytometry); ③ Serological detection of EBV antibodies indicating any of the following: positive anti-VCA-IgM; positive anti-EA-IgG; or simultaneous positivity for anti-VCA-IgM, anti-VCA-IgG, and anti-EBNA-IgG.
   3. At least one evaluable lymphoma lesion according to Lugano criteria, or confirmed active lytic EBV infection.
3. Performance Status: ECOG score 0-2 and expected survival ≥3 months;
4. Age: 18-70 years, regardless of sex;
5. Hematologic Criteria:

   * Absolute neutrophil count (ANC) ≥1.0×10⁹/L;
   * Hemoglobin >60 g/L;
   * CD3+ T-cell count >0.5×10⁹/L;
   * Platelet count >30×10⁹/L;
6. Organ Function:

   * Creatinine clearance ≥60 mL/min;
   * ALT/AST ≤2× upper limit of normal (ULN);
   * Total bilirubin ≤2× ULN;
   * Left ventricular ejection fraction (LVEF) ≥50%, no pericardial effusion, and no clinically significant ECG abnormalities;
   * Minimal or no pleural/ascitic fluid;
   * Oxygen saturation ≥95%;
7. Contraception:

   * Women of childbearing potential must have a negative pregnancy test and agree to use effective contraception until the last follow-up;
   * Male participants with fertile partners must agree to use effective contraception until the last follow-up;
8. Informed Consent: Psychologically stable, capable of understanding the study's purpose and procedures, willing to participate voluntarily, and able to provide signed informed consent and comply with protocol requirements.

Exclusion Criteria:

1. Active Infections: Presence of active hepatitis A, B, or C infection, or other uncontrolled severe active infections (excluding EBV infection);
2. Immunosuppression:

   * History of acquired immunodeficiency syndrome (AIDS);
   * Chronic use of immunosuppressants (including corticosteroids at doses equivalent to >15 mg/day of prednisone) for other conditions;
3. Cardiac Dysfunction:

   1. NYHA Class III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass grafting within the past 6 months;
   3. Clinically significant ventricular arrhythmia or unexplained syncope;
   4. History of severe non-ischemic cardiomyopathy;
   5. Cardiac insufficiency (left ventricular ejection fraction <45%) within 8 weeks prior to apheresis;
4. Pregnancy/Contraception:

   * Pregnant or lactating women;
   * Participants (male or female) unwilling to use contraception;
5. Hepatic/Renal Impairment:

   * AST/ALT >3× upper limit of normal (ULN);
   * Total bilirubin >3× ULN;
   * Creatinine clearance <60 mL/min;
6. Allergies: History of severe hypersensitivity to any study drugs;
7. Prior Stem Cell Transplant: Must have discontinued immunosuppressants for >6 weeks post-transplant with no signs of graft-versus-host disease (GVHD);
8. Other Exclusionary Conditions: Any other condition deemed unsuitable by the investigator (e.g., coagulation disorders, hemolytic anemia, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2030-11-10 (Estimated); Study Completion 2032-11-20 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Month 12 post CAR-T infusion
  The percentage of patients with complete response (CR) and partial response (PR) according to the RECIL 2017 criteria determined by the study investigators
EBV DNA clearance rate | Month 12 post CAR-T infusion
  Defined as the proportion of patients achieving two consecutive negative tests in plasma or whole blood at least 7 days apart following treatment, relative to the total treated population
Treatment Emergent Adverse Event (TEAE) | Within 3 months post-infusion
  TEAE is defined as an adverse event that occurs or worsens after receiving the first dose of the trial drug

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 1 yesr post CAR-T infusion
  PFS is defined as the time from the GP350 CAR-T infusion date to the date of disease progression
Overall Survival (OS) | 1 yesr post CAR-T infusion
  OS is the time from date of GP350 CAR-T infusion to the date of death due to any reason

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No